CLINICAL TRIAL: NCT01895231
Title: A Randomized, Prospective, Double-Blind, Comparative Placebo-Controlled Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by Infusions to Iron-Deficient Blood Donors
Brief Title: A Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by Infusions to Iron-deficient Blood Donors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: Max Neeman (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-Monofer-BD-02
Record Dates: First submitted 2013-06-26; First posted 2013-07-10 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — iron isomaltoside 1000; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron isomaltoside 1000 (Experimental): Monofer® 1000 mg IV infusion over 15 minutes
  Interventions: Drug: Iron isomaltoside 1000 (Monofer®)
- Placebo (Placebo Comparator): 0.9 % saline Infusion over 15 min
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iron isomaltoside 1000 (Monofer®)
  Other Names: Monofer®
  Arms: Iron isomaltoside 1000
Drug: Placebo
  Other Names: 0.9 % saline
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the effect of IV iron isomaltoside 1000 compared with placebo on Hb in first-time female donors with p-ferritin below 30 µg/L

DETAILED DESCRIPTION:
At present, clinical efficacy and safety data is available for iron isomaltoside 1000 administered to patients with IDA requiring iron therapy. However, there is a need for clinical efficacy and safety data within iron deficiency without anaemia which is e.g. observed in blood donors. Thus, this study is planned to compare the efficacy and safety of parenteral iron isomaltoside 1000 with placebo in female blood donors with a p-ferritin below 30 µg/L.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥ 18 years
2. First-time donor
3. P-ferritin < 30 µg/L
4. Willingness to participate and signed the informed consent form

Exclusion Criteria:

1. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and haemosiderosis)
2. Known hypersensitivity to any excipients in the investigational drug products
3. History of drug related allergies
4. History of severe asthma
5. Decompensated liver cirrhosis and hepatitis (defined as ALAT > 3 times upper limit of normal)
6. Active acute or chronic infections (assessed by clinical judgement supplied with White Blood Cells (WBC) and C-Reactive Protein (CRP))
7. Rheumatoid arthritis with symptoms or signs of active inflammation
8. Subjects who are pregnant or nursing. In order to avoid pregnancy, women have to be postmenopausal (at least 12 months since last menstruation), surgically sterile, or use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product: intrauterine devices and hormonal contraceptives (contraceptive pills, implants, transdermal patches, vaginal devices, or hormonal injections with prolonged release)
9. Participation in any other clinical study where the study drug has not passed 5 half-lives prior to the screening
10. Untreated vitamin B12 or folate deficiency
11. Treated with other IV or oral iron products within 4 weeks prior to the screening
12. Treated with Erythropoietin (EPO) within 4 weeks prior to the screening
13. Any other medical condition that, in the opinion of the Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Hb concentration | From baseline and until t= 6 months
  The primary endpoint is to measure and compare the change in Hb concentration from baseline to right before the third blood donation in the two study arms

SECONDARY OUTCOMES:
Change in Hb concentration | From baseline and until t=3 months
  Change in Hb concentrations from baseline to right before second donation
Ability to complete 3 blood donations | From baseline and until t=6 months
  Number of subjects who cannot complete three donations due to low Hb
Change in p-iron | From baseline and until week 12
Change in fatigue symptoms | From baseline and until week 12
Exercise tolerance | From baseline to week 3
  Change in exercise tolerance from baseline to 3 weeks after baseline measured by a two-step test on bike
Number of adverse drug reactions | From screening and until t= 6 months
Change in p-ferritin | From baseline and until week 12
Change in Transferrin Saturation (TSAT) | From baseline until week 12
Change in reticulocyte count | From Baseline to week 12
Change in haematology parameters | From baseline and until t= 6 months
Change in RLS symptoms | From baseline and until t= 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nørgaard, Principal Investigator — RH Blodbanken
Locations (1):
- Copenhagen, Denmark